CLINICAL TRIAL: NCT02501122
Title: Cost Savings From Non-pharmacological Interventions for Pediatric Patients Undergoing Diagnostic Imaging at Nationwide Children's Hospital
Brief Title: Retrospective Analysis in Quality of Care Measures in Pediatric Adenotonsillectomy Patients
Status: Completed | Type: Observational
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB 15-00264
Record Dates: First submitted 2015-05-20; First posted 2015-07-17 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Adenotonsillectomy
Keywords: Quality; hospital care; adenotonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adenotonsillectomy: Measuring quality of care in patients undergoing adenotonsillectomy.
  Interventions: Other: Pediatric Health Information System (PHIS), Partners for Kids (PFK) and Nationwide Children's Hospital Perioperative Database

INTERVENTIONS:
Other: Pediatric Health Information System (PHIS), Partners for Kids (PFK) and Nationwide Children's Hospital Perioperative Database — Utilizing these databases to assess standards for quality of care measures in adenotonsillectomy patients.

SUMMARY:
The purpose of this study is to interrogate the Partners for Kids (PFK) and the pediatric health information (PHIS) databases in addition to our own perioperative Nationwide Children's data base to look at outcomes, resource utilization, and cost trends for adenotonsillectomy in the nationally versus locally. The investigators also want compare Nationwide Children's to other regional and national tertiary pediatric institutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergone an adenotonsillectomy, tonsillectomy or adenoidectomy during the past 2 years (2013-2015) who have ICD-9 codes (International Classification of Diseases) in the databases

Exclusion Criteria:

* Non-adenotonsillectomy patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone anesthesia for adenotonsillectomy, tonsillectomy or adenoidectomy during 2013-2015 at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gather data from PHIS and contrast local databases (PFK versus Nationwide Children's) | after patient's discharge, an expected average between 6 months to 2 years
  The significance is to identify outcome measures, resource utilization, and cost of adenotonsillectomy nationally as well as locally.

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Raman, MD, Principal Investigator — Nationwide Children's Hospital